CLINICAL TRIAL: NCT00826202
Title: D-Serine vs Placebo for the Schizophrenia Prodrome
Brief Title: D-serine for the Schizophrenia Prodrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Yale University (Other); The Zucker Hillside Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08I/C33; CDDG 1 U01 MH074356-01
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia Prodrome
Keywords: schizophrenia; d-serine; prodrome
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D serine (Experimental): 60 mg/kg/day
  Interventions: Drug: D-serine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-serine — 60 mg/kg/day
  Arms: D serine
Other: Placebo — Inert Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the safety and efficacy of D-serine as an early intervention treatment for the schizophrenia prodrome condition. This study is a placebo-controlled trial of D-serine in the symptomatic treatment of patients with the schizophrenia prodrome. Seventy two subjects meeting criteria for the schizophrenia prodrome will be included in this study, 24 at each site (Yale, Nathan Kline Institute and Zucker Hillside Hospital). The primary outcome measures will include symptom and neuropsychological measures. The duration of this study is two and a half years.

This research with D-serine holds out the prospect of direct benefit for the patient's current symptoms. Subjects may also benefit from the close monitoring of their symptoms, so that, if schizophrenic psychosis does occur, the psychosis will be recognized and treatment may begin with minimal delay. This study also could be of benefit by suggesting a promising lead in early intervention in the schizophrenic prodrome.

Overall Design Summary. We propose for prodromal patients to be randomized to D-serine vs placebo for 16 weeks. To insure that all subjects have the opportunity to receive D-serine, there will be an optional 16 week cross-over trial on the alternate study medication. No subject will be on D-serine for longer than 16 weeks. Admission criteria, Assessment Procedures, and Study Design will be the same across all sites. The procedures and timeline are shown in Table 1. The procedures and timeline are the same for the initial randomized 16 week trial and the optional cross-over trial on the alternate study medication. If patient's opt for the 16 week treatment on the alternate medication, we will use their assessments from end of initial treatment as baseline for 16 week treatment on alternate medication. Subjects will be seen for two preliminary visits, then once in treatment, subjects will be seen weekly for the first 5 visits then biweekly thereafter. A safety blood and urine collection will be done on day 3 (3 days after the start of study medication). Vital signs and weight, blood draw and urine collection for safety measures, urine pregnancy test and urine for toxicology will be repeated throughout treatment. Adverse effects ratings and symptom assessments will be repeated at each visit. Neuropsychological assessment and optional "Biomarker study" visual, auditory and ERPs tasks will be administered during one of the two preliminary visits then again at study endpoint. Any patients who convert to frank psychosis will be referred/offered immediate treatment.

ELIGIBILITY:
Inclusion criteria:

1. treatment seeking subjects ages 13-35 who meet criteria for the schizophrenia prodrome (see criteria below) and who are able to give written informed assent or consent.
2. Subjects must score at least 20 on the Scale of Prodromal Symptoms (SOPS) total score at visit -1.
3. Patients may be receiving ongoing treatment with antipsychotic, antidepressant or anti-anxiety medications as prescribed by their treating physician, or may be medication free.
4. Patients may enroll in the treatment phase only if they have been on fixed medication dosage for at least 4 weeks. If possible, medication will be held constant during course of study. Subjects will not be excluded or dropped from the study if they have a psychiatric diagnosis or must start a new medication unless the diagnosis is "psychosis". Medication changes and increases or decreases in medication will be permitted at the discretion of the treating physician, and, if they occur, will be treated as secondary outcome measures.

Exclusion criteria:

1. inability to give informed assent or consent,
2. history of psychosis (e.g. frank delusions, hallucinations, or thought disorder),
3. psychotropic medication begun or dose adjusted within 4 weeks of visit 0,
4. contraindication to study medication,
5. inclusion symptoms better accounted for by comorbid diagnosis,
6. treatment need for comorbid diagnosis outweighs that for prodromal symptoms,
7. unstable medical illness,
8. females who are of childbearing potential but are not taking adequate contraceptive precautions or who are pregnant or breast feeding,
9. alcohol or drug abuse or dependence in the past three months,
10. either of the following: Subjects with significant renal disease or estimated GFR below 60 (MDRD, http://www.kidney.org/professionals/kdoqi/gfr_calculator.cfm) will be excluded (see below for details). Any subject taking or unwilling to avoid other nephrotoxic agents during the course of the study (NSAIDS, ACE inhibitors, ARB's, calcineurin inhibitors, or aminoglycosides) will also be excluded. Therefore, patients will be asked during the study to take acetaminophen (e.g. if they have a headache) and to avoid taking ibuprofen.

For adolescents (ages 13-17), more stringent renal exclusion criteria will be adhered to:

1. estimated GFR is < 89 cc/min/1.73 m2 as calculated by the Schwartz formula (http://www.kidney.org/professionals/kdoqi/gfr_calculatorPed.cfm),
2. difference of ≥0.3mg/dl between the two baseline serum creatinine values,
3. baseline proteinuria defined by a spot urine protein:creatinine of 0.2 or greater, or
4. baseline glucosuria (the presence of glucosuria).

Schizophrenia Prodrome Criteria:

We will be enrolling both Attenuated Positive Syndrome (APS) [1], Genetic Familial Risk (GFR) [1] and Clinically High Risk Negative (CHR-) symptom prodromes to this study. A separate analysis will be done for the APS and CHR- patients.

1. Attenuated Positive Syndrome: One or more of the 5 SOPS positive items scoring in the prodromal range (rating of 3-5) AND Symptoms beginning within the past year or increasing 1 or more points within the past year AND Symptoms occurring at least once per wk for last month.
2. Genetic Familial Risk: First degree relative with history of any psychotic disorder OR Criteria for schizotypal personality disorder met in patient AND GAF drop of at least 30% over the last month vs 1 year ago. In our experience, very few patients only meet criteria for this syndrome.
3. CHR-: To make criteria, social isolation must be present along with either flat affect or impairment in the occupational role. Therefore to meet criteria for CHR-, Social Anhedonia (N1) has to be present at a score of 3 or above, and, in addition, one of the other two symptoms (N3 or N6) listed must also present at a minimum level of 3. Note: a score of "6" on these items is not considered exclusionary.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Javitt, MD, PhD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Zucker Hillside Hospital, Glen Oaks, New York
  - New York State Psychiatric Institute, New York, New York
  - Nathan Kline Institute, Orangeburg, New York

REFERENCES:
- [Result] Kantrowitz JT, Woods SW, Petkova E, Cornblatt B, Corcoran CM, Chen H, Silipo G, Javitt DC. D-serine for the treatment of negative symptoms in individuals at clinical high risk of schizophrenia: a pilot, double-blind, placebo-controlled, randomised parallel group mechanistic proof-of-concept trial. Lancet Psychiatry. 2015 May;2(5):403-412. doi: 10.1016/S2215-0366(15)00098-X. Epub 2015 Apr 28. PMID 26360284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D Serine | Placebo
Started | 20 | 24
Completed Visit 4 (1st Efficacy Visit) | 15 | 20
Completed | 10 | 11
Not Completed | 10 | 13

BASELINE CHARACTERISTICS:
Population: Includes 35 subjects who received at least one post-baseline efficacy evaluation
Groups:
- Total: Total of all reporting groups
Arm/Group | D Serine | Placebo | Total
Number analyzed (Participants) | 15 | 20 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 9 | 16
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (4.9) | 19 (3.5) | 19.5 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 8 | 15 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 20 | 35

OUTCOME MEASURES:

1. Secondary Outcome: Scale of Prodromal Symptoms (SOPS) Total
Description: The SOPS Total consists of five Positive Symptom items, six Negative Symptom items, four Disorganization Symptom items, and four General Symptom items. Each item has a severity scale rating from 0 (Never, Absent) to 6 (Severe/Extreme-and Psychotic, for the positive items). The severity of the prodromal state is judged according to the sum of the ratings from each of the SOPS items and ranges from 0 to 114.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D Serine | Placebo
Number analyzed (Participants) | 15 | 20
units on a scale | 23.9 (2.8) | 30.5 (2.4)
Statistical Analysis 1: Comparison: D Serine vs Placebo; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis; cohen's d= 0.67

2. Secondary Outcome: IL6 Levels
Description: Final IL6 levels (pg/ml) in available subjects
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: final IL6 level (pg/ml))
Arm/Group | D Serine | Placebo
Number analyzed (Participants) | 11 | 16
final IL6 level (pg/ml)) | .49 (.25) | .79 (.52)
Statistical Analysis 1: Comparison: D Serine vs Placebo; Test type: Superiority or Other; p = .056, t-test, 2 sided; cohen's d=0.84

3. Primary Outcome: Scale of Prodromal Symptoms (SOPS) Negative Scale
Description: The SOPS Negative symptom scale consists of six Negative Symptom items. Each item has a severity scale rating from 0 (Never, Absent) to 6 (Severe/Extreme). The severity of the prodromal state is judged according to the sum of the ratings from each of the SOPS items and ranges from 0 to 36.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: SOPS negative final score
Arm/Group | D Serine | Placebo
Number analyzed (Participants) | 15 | 20
SOPS negative final score | 7.6 (1.4) | 11.3 (1.2)
Statistical Analysis 1: Comparison: D Serine vs Placebo; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis; Cohen's d=0.68

4. Secondary Outcome: Pittsburgh Sleep Quality Index Score
Description: The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and five questions rated by the bed partner or roommate. The latter five questions are used for clinical information only, are not tabulated in the scoring of the PSQI. The 19 self-rated questions assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep-related problems. These I9 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores
Time Frame: 16 weeks
Population: Completers at NYSPI and NKI sites
Measure: Mean (Standard Deviation); unit: final score
Arm/Group | D Serine | Placebo
Number analyzed (Participants) | 8 | 11
final score | 4 (2.9) | 7.7 (3.5)
Statistical Analysis 1: Comparison: D Serine vs Placebo; Test type: Superiority or Other; p = 0.12, Mixed Models Analysis; cohen's d=0.93

ADVERSE EVENTS:
Arm/Group | D Serine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/24
Other Adverse Events (participants affected / at risk) | 2/20 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D Serine (N=20) | Placebo (N=24)
suicidal thoughts-hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — patient remained in study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D Serine (N=20) | Placebo (N=24)
Out of range renal values (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No